CLINICAL TRIAL: NCT04014543
Title: Assessing the Quality of Life of Caregivers and Before and After the Position of Gastronomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-65; 2018-A03284-51 (Registry Identifier: ANSM)
Record Dates: First submitted 2019-06-18; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Gastrostomy
MeSH Terms: interventions — Contact Tracing

STUDY DESIGN:
Intervention Model Description: caregivers and children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastrostomy (Experimental): Gastrostomy involves creating an opening between the skin and the stomach. It allows the administration of nutrition solutes or food directly into the stomach without passing through the mouth and esophagus. It is a method widely used since the 1980s for enteral nutrition.
  In the field of pediatrics, gastrostomy is considered in chronic diseases when enteral nutrition is necessary in the long term.
  Interventions: Other: gastronomy

INTERVENTIONS:
Other: gastronomy — to study the quality of life of caregivers and children with generic questionnaires (13-16), validated and used in other pathologies and chronic diseases of the child.
  This will allow reproducibility and comparisons to other populations, general or other chronic diseases (acute leukemias ...) This is to conduct a pilot study, preliminary to the construction of a larger study, longitudinal with several evaluation times.
  Other Names: investigation

SUMMARY:
The goal of this reasearch project is to study the quality of life of caregivers and children with generic questionnaires, validated and used in other pathologies and chronic diseases of the child.

This will allow reproducibility and comparisons to other populations, general or other chronic diseases (acute leukemias ...) This is to conduct a pilot study, preliminary to the construction of a larger study, longitudinal with several evaluation times.

DETAILED DESCRIPTION:
Gastrostomy involves creating an opening between the skin and the stomach. It allows the administration of nutrition solutes or food directly into the stomach without passing through the mouth and esophagus. It is a method widely used since the 1980s for enteral nutrition.

In the field of pediatrics, gastrostomy is considered in chronic diseases when enteral nutrition is necessary in the long term. It allows weight gain and improves nutritional status. The percutaneous endoscopic method is nowadays one of the most widespread methods that has proven effective on growth and nutrition, with few side effects .

Few studies have analyzed children's quality of life after gastrostomy. On the one hand, it increases the perceived health of the child after the placement of the caregiver's point of view. It allows a reduction of the stress of the parents, at a distance from the pose, and its insertion would be chosen again by the parents if it were to do again. Meals and medication administration would be easier for parents. But on the other hand, its insertion is often difficult for families to experience, on the one hand by changing the diet . The family dynamics are modified and it would lead to logistical constraints for meals or outings. The vision of the body diagram would also be altered. Following a systematic review of the literature conducted in early 2018, there are currently only 7 longitudinal prospective studies assessing the quality of life of caregivers before and after gastrostomy. No study is French. The numbers are relatively small. All of these studies assess the quality of life of caregivers only, without assessing the quality of life of the child due to age-related constraints and causal pathology. Six of seven studies show an improvement in the quality of life of caregivers after the pose. The 7th study, which is the only multicentre study, shows no improvement in the quality of life, with an increase in time for care and cost. This is a US study in 3 centers comparing 50 children with and without gastrostomy at 3 assessment points at 0, 3 and 6 months. Children with gastrostomy would require more time for care and a cost. This study found no improvement in caregivers' quality of life and mood on a depression scale. However, the 2 groups were not similar in terms of pathology with more hematological pathologies and fewer degenerative neurological pathologies in the group without gastrostomy. The care, devices and materials are paid in the US which is not the case in France and should not impact on the quality of life. These studies, with the exception of 2 who used the SF-36 questionnaire, were conducted with different and non-standardized self-questionnaires.

None of these studies conducted a direct assessment of the child using a questionnaire designed for them. This assessment of children can be performed in children of understanding age and having a pathology that allows them to communicate. It allows an approach and a direct vision of the quality of life. The quality of life of the siblings has also not been studied in these studies whereas it is impacted in the chronic diseases in the brothers and sisters. Our goal is to study the quality of life of caregivers and children with generic questionnaires, validated and used in other pathologies and chronic diseases of the child. This will allow reproducibility and comparisons to other populations, general or other chronic diseases (acute leukemias ...) This is to conduct a pilot study, preliminary to the construction of a larger study, longitudinal with several evaluation times.

ELIGIBILITY:
Inclusion Criteria:

Child:

* 1 month to 17 years old;
* Accepting to participate in the study;
* Having a pathology requiring enteral nutrition in the long term exclusive or mixed;
* Having the programming of the insertion of percutaneous gastrostomy in the multidisciplinary pediatric ward.

Helping :

* Parent or representative of the parental authority of a child meeting the inclusion criteria above;
* Accepting to participate in the study;
* Having the ability to comply with the protocol requirements (in particular: understanding and speaking French).
* Siblings:
* 8 to 17 years old;
* Accepting to participate in the study;
* Having the ability to comply with the requirements of the protocol (understanding and speaking French, presenting no sensory, motor, cognitive or severe chronic illness);
* Living in the same home as the sick child.

Exclusion Criteria:

Child:

* Refusing to participate in the study;
* Surgical, radiological or emergency gastrostomy.

Helping :

* Inability to comply with study protocol, or investigator uncertainty about willingness or ability to comply with protocol requirements;
* Refusing to participate in the study.
* Siblings:
* Refusing to participate in the study.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the body mass index | 19 moths
  Observation of a decrease in body mass index after gastrostomy

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France